CLINICAL TRIAL: NCT07227558
Title: Improving Information Sharing Between Family Caregivers and Home Care Aides Caring for Persons Living With ADRD
Brief Title: Improving Information Sharing Between Family Caregivers and Home Care Aides
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00022916; 5K01AG080079-03 (NIH)
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Shared Care
Keywords: Shared Care; Family Caregiving; Paid Caregiving

STUDY DESIGN:
Intervention Model Description: The interventional study model will include a home care role and preference guide to improve information sharing and clarify role expectations between family caregivers and home care aides of older adults with disabilities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GRACE (Other): Role and preference guide for family caregivers and home care aides
  Interventions: Other: GRACE

INTERVENTIONS:
Other: GRACE — GRACE- Guide for Role Awareness and Care Engagement is a role and preference guide designed to improve information sharing and clarify role expectations between family caregivers and home care aides of older adults. This guide will outline the various domains of providing care services and preferences for older adults such as daily routine and preferred activities. The intervention will be delivered in-person to the family caregiver and home care aide at the care recipient's home.

SUMMARY:
This study will assess the feasibility and acceptability of delivering a home care role and preference guide to up to 50 family caregivers and home care aides of persons living with disability for the purpose of identifying roles between family caregivers and home care aides.

DETAILED DESCRIPTION:
This study will assess the feasibility and acceptability of delivering a home care role and preference guide to family caregivers and home care aides of persons living with disability for the purpose of identifying roles between family caregivers and home care aides, as well as preliminary effects on older adult social engagement, caregiver distress, continuity, and feelings of being overwhelmed, family caregiver/direct care worker preparedness, relational coordination, and service satisfaction. The intervention will involve delivering the home care role and preference guide to up to 50 family caregiver-home care care aide dyads to demonstrate the feasibility of collecting primary endpoints relating to older adults' outcomes to be examined in a future ePCT as well as intervention acceptability. Information about family caregivers and home care aide perspectives will be collected at enrollment, 2- and 4-weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Home care agency aide:

   * English speaking,
   * home care aides, personal care aides, or personal care aides, providing services to older adults with ADRD.
2. Family or unpaid caregiver eligible for the study if:

   * 18 years and older
   * English speaking
   * hear well enough to communicate by telephone
   * identify themselves as the primary family member or unpaid (friend/companion) caregiver

Exclusion Criteria:

1. Home care aides are ineligible if:

   * non-English speaking
   * certified nursing assistants, nursing assistant, home health aides, or medication technicians.
2. Family/unpaid caregivers ineligible if:

   * less than 18 years old
   * non-English speaking
   * do not hear well enough to communicate by telephone
   * two or more incorrect answers or not being able to respond to a validated 6-item telephone screening instrument
   * are not identified as the person's primary caregiver, or are paid for services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability as assessed by survey | 2 week and 4 weeks
  Participants will be asked to rate their overall feedback of the role and preference guide. Participants will be asked how often they used the guide since the last study time point using a scale from 1 to 5 (1=Never, 2=Rarely, 3=Occasionally, 4= Often, 5 Constantly) where higher scores indicate greater frequency of use.
Feasibility as assessed by survey | 2 week and 4 weeks
  Participants will be asked about how helpful the guide was using a scale from 1 to 5:1=Not helpful at all, 2=Not too helpful, 3=Somewhat helpful, 4=Pretty helpful, 5=Very helpful, where higher scores indicate more helpful. More affirmative responses indicate better feasibility of the guide.
Low Social Engagement as assessed by survey question | Baseline, 2 weeks and 4 weeks
  Low social engagement measures an older adult's ability to participate in social activities of longstanding interest reported by the caregiver. This item is measured on a scale from 0-3 (0=Occurred in the last 3 days, 1=Occurred within the last week, 2=Occurred within the last month, 3=Last occurred more than one month ago) where higher scores mean lesser ability to participate in social activities.
Caregiver is Overwhelmed as assessed by survey question | Baseline, 2 weeks and 4 weeks
  Caregivers' feelings of being overwhelmed measures how often a caregiver is overwhelmed by aspects of caregiving responsibilities and older adults' illness. This item is measured using a scale from 1-5 (1=Never, 2=Rarely, 3=Occasionally, 4=Often, 5= Constantly) where higher scores mean greater feelings of being overwhelmed.
Caregiver Distress assessed by survey question | Baseline, 2 weeks and 4 weeks
  Caregivers' feelings of distress measures how often a caregiver is distressed by aspects of caregiving responsibilities and older adults' illness. This item is measured using a scale from 1-5 (1=Never, 2=Rarely, 3=Occasionally, 4=Often, 5= Constantly) where higher scores mean greater feelings of distress.
Caregiver Continuity assessed by survey item | Baseline, 2 weeks and 4 weeks
  Caregivers continuity measures how feelings on inability to continue caregiving. This item is measured using a scale from 1-5 (1=Never, 2=Rarely, 3=Occasionally, 4=Often, 5= Constantly) where higher scores mean greater feelings of distress.
Caregiver Preparedness assessed by The Caregiving Preparedness Scale (CPS) | Baseline, 2 weeks and 4 weeks
  The Caregiving Preparedness Scale (CPS) is an 8-item uni-dimensional instrument that evaluates the extent to which a caregiver and direct care worker feels prepared to meet the psychological and physical needs of a patient (client). The scale was originally developed for family caregivers and has been used to assess caregiver preparedness in direct care workers in prior work. Responses are categorized with a 5-level likert scale: Not at all prepared; not too prepared; somewhat well prepared; pretty well prepared; very well prepared. The total scale score, which is a mean of all items scores, ranges between 0 and 4 with higher score indicating better preparedness.
Relational Coordination assessed by survey | Baseline, 2 weeks and 4 weeks
  Relational coordination suggests that effective coordination occurs through frequent, high-quality communication that is supported by relationships of shared goals, shared knowledge, and mutual respect. Its measurement has been applied across several settings, including home care.
  Family caregivers and direct care workers will rate interactions with each other along three dimensions, with seven questions on a five-point scale related to the components of relational coordination. Four items related to communication include: frequency, timeliness, accuracy, and problem-solving. Three items measured relationships: shared knowledge, goals, and respect for each other. The mean of each of the seven items is calculated for each group (family caregivers and direct care workers). The total score for all items ranges from 7 to 35 where higher scores indicate better coordination and communication among family caregiver and direct care worker.
Direct Care Worker Job Satisfaction assessed by survey question | Baseline, 2 weeks and 4 weeks
  Job satisfaction measures the direct care worker's overall job satisfaction on a scale from 1-4 (1= Very dissatisfied, 2=Dissatisfied, 3=Satisfied, 4=Very Satisfied). Higher score is better.
Number of participants with new Direct Care Worker | 2 weeks and 4 weeks
  Direct Care Worker Turnover measure changes in the enrolled direct care worker participant in the study from the time baseline is completed to study endpoint at 4 weeks. Caregivers will be asked if the direct care worker left and at what time point in the study, and if the participant was assigned or hired a new worker. This will be measured using affirmative responses (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Chanee Fabius, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health